CLINICAL TRIAL: NCT06241560
Title: An Open-label, Single-group Trial to Evaluate the Effect of Pirfenidone on the Pharmacokinetics of a Single Oral Dose of BI 1015550
Brief Title: A Study in People With Idiopathic Pulmonary Fibrosis to Test Whether Pirfenidone Influences the Amount of BI 1015550 in the Blood
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1305-0035
Record Dates: First submitted 2024-01-29; First posted 2024-02-05 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — BI 1015550; pirfenidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BI 1015550, then Pirfenidone + BI 1015550 (Experimental)
  Interventions: Drug: BI 1015550; Drug: Pirfenidone

INTERVENTIONS:
Drug: BI 1015550 — BI 1015550
  Other Names: Nerandomilast, JASCAYD®
Drug: Pirfenidone — Pirfenidone
  Other Names: Esbriet

SUMMARY:
This study is open to adults with idiopathic pulmonary fibrosis (IPF) who are 40 years and older. The purpose of this study is to find out whether a medicine called pirfenidone changes the amount of a medicine called BI 1015550 in the blood. Some people may take more than one medicine at a time. Therefore, it is important to understand how different medicines influence one another.

Participants take one dose of BI 1015550 as a tablet. Participants then take one tablet of pirfenidone 3 times a day for one week. The dose is then increased to 2 tablets 3 times a day for the second week. In the third week the dose is increased further to 3 tablets 3 times a day. Participants then take another dose of BI 1015550 as a tablet.

Participants are in the study for a little over 1 month. During this time, they visit the study site 15 times. Two of the visits include overnight stays at the study site. The study staff also contacts the participants by phone. During the visits, the doctors collect information about participants' health and take blood samples from the participants. They compare the amount of pirfenidone and BI 1015550 in the blood. Doctors also regularly check participants' health and take note of any unwanted effects.

ELIGIBILITY:
Inclusion criteria:

* Male or female patients aged ≥40 years old at the time of signed consent
* Patients with idiopathic pulmonary fibrosis (IPF) and an indication/no contraindication for treatment with pirfenidone based on investigator's judgement.
* Body mass index (BMI) of 18.5 to 29.9 kg/m^2 (inclusive)
* Signed and dated written informed consent in accordance with International Conference of Harmonization-Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial
* Women of childbearing potential (WOCBP) must be ready and able to use highly effective methods of birth control. WOCBP taking oral contraceptives (OC) also have to use one barrier method

Exclusion criteria:

* Patients with a significant disease or condition other than IPF, which in the opinion of the investigator, may put the patient at risk because of participation, interfere with study procedures, or cause concern regarding the patient's ability to participate in the study
* Acute IPF exacerbation within 1 month prior to Visit 1 and/or during the screening period (investigator-determined).
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >2.5 x ULN or total Bilirubin >1.5 x upper limit of normal (ULN) at Visit 1
* Patients with underlying liver cirrhosis (Child Pugh A, B or C hepatic impairment)
* Cardiovascular diseases, any of the following:

  * Severe hypertension (uncontrolled under treatment ≥160/100 mmHg at multiple occasions) within 3 months of Visit 1
  * Myocardial infarction, stroke or transient ischemic attack within 6 months of Visit 1
  * Unstable cardiac angina within 6 months of Visit 1
* Chronic kidney disease with estimated glomerular filtration rate (eGFR) less than 90 ml/min/1.73 m^2 at Visit 1/screening (Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] formula or Japanese version of CKD-EPI for Japanese patients)
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
* Relevant chronic or acute infections including but not limited to human immunodeficiency virus (HIV) and viral hepatitis
* Further exclusion criteria apply

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-03-13 (Estimated); Primary Completion 2026-08-04 (Estimated); Study Completion 2026-08-06 (Estimated)

PRIMARY OUTCOMES:
Area under the concentration-time curve of BI 1015550 in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz) | Up to day 34
Maximum measured concentration of BI 1015550 in plasma (Cmax) | Up to day 34

SECONDARY OUTCOMES:
Area under the concentration-time curve of BI 1015550 in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) | Up to day 34

CONTACTS AND LOCATIONS:
Locations (3):
- Renovatio Clinical-The Woodlands-69551, The Woodlands, Texas, United States
- Georgia (2):
  - LTD The First Medical Center, Tbilisi
  - LTD "Aversi clinic", Tbilisi

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization). For more details refer to: https://www.clinicalstudies.boehringer-ingelheim.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.clinicalstudies.boehringer-ingelheim.com/msw/datasharing